CLINICAL TRIAL: NCT04023227
Title: A Multicenter, Prospective, Randomized, Open-label, Blinded-endpoint, Phase 4 Study to Evaluate the Efficacy and Safety of Sacubitril/Valsartan Compared With Enalapril on Morbidity, Mortality, and NT-proBNP Change in Patients With Chronic Chagas' Cardiomyopathy. The Study is Also Know as Prevention And Reduction of Adverse Outcomes in Chagasic Heart failUre Trial Evaluation (PARACHUTE-HF).
Brief Title: Efficacy and Safety of Sacubitril/Valsartan Compared With Enalapril on Morbidity, Mortality, and NT-proBNP Change in Patients With CCC
Acronym: PARACHUTE-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLCZ696B3302
Record Dates: First submitted 2019-07-10; First posted 2019-07-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chagas Disease; Heart Failure
Keywords: Chagas' disease; heart failure; angiotensin receptor-neprilysin inhibitor; ARNI; ARB; ACEI; sacubitril/valsartan; enalapril
MeSH Terms: conditions — Chagas Disease; Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Enalapril

STUDY DESIGN:
Intervention Model Description: This is a Phase 4, multinational, multicenter, parallel-group, prospective, randomized, open-label, blinded-endpoint adjudication, active-controlled study to demonstrate superiority of sacubitril/valsartan over enalapril in improving a composite of CV events (CV death or first HF hospitalization), or in causing greater reduction or lesser increase in NT-proBNP levels at Week 12 in participants with HFrEF caused by CCC.
Who Masked: Outcomes Assessor
Masking Description: Endpoint Adjudication Committee will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacubitril/valsartan (Experimental): Sacubitril/valsartan 200 mg b.i.d.
  Following randomization, patients will receive sacubitril/valsartan in titrated doses from level 1 up to level 3 (50, 100 and 200 mg twice daily).
  Participants taking ACEIs who are randomized to sacubitril/valsartan will do a 36-hour ACEI washout before they start taking the study drug
  Sacubitril/valsartan in dose levels of 50 mg, 100 mg, and 200 mg are equivalent to sacubitril/valsartan 24/26 mg, 49/51 mg and 97/103 mg, respectively
  Interventions: Drug: Sacubitril/valsartan
- Enalapril (Active Comparator): Enalapril 10 mg b.i.d.
  Following randomization, patients will receive the enalapril in titrated doses from level 1 up to level 3 (2.5, 5 and 10 mg twice daily).
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Sacubitril/valsartan — 50 (24/26) mg, 100 (49/51) mg and 200 (97/103) mg will be available for dose adjustments.
  Other Names: LCZ696; Entresto; Vymada
  Arms: Sacubitril/valsartan
Drug: Enalapril — 5 mg and 10 mg will be available for dose adjustments.
  Other Names: Renitec
  Arms: Enalapril

SUMMARY:
The purpose of this study is to evaluate the effect of sacubitril/valsartan 200 mg BID compared with enalapril 10 mg BID, in addition to conventional heart failure (HF) treatment, in improving a hierarchical composite of cardiovascular (CV) events (i.e. CV death or the occurrence of first HF hospitalization) and causing a greater reduction in n terminal prohormone of brain natriuretic peptide (NT-proBNP, at Week 12 from Baseline) in participants with HF with reduced ejection fraction (HFrEF) caused by CCC.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female ≥ 18 years of age
* Diagnosis of NYHA Class II-IV HFrEF established by:

  1. LVEF ≤ 40% within 12 months prior to Visit 1 made by any local measurement using echocardiography, multiple gated acquisition scan (MUGA), computerized tomography (CT) scanning, magnetic resonance imaging (MRI), or ventricular angiography, provided no subsequent measurement above 40% AND
  2. NT-proBNP ≥ 600 pg/mL (or BNP ≥ 150 pg/mL) at Visit 1 OR
  3. NT-proBNP ≥ 400 pg/mL (or BNP ≥ 100 pg/mL) at Visit 1 and a hospitalization for HF within the last 12 months
* Chagas' disease diagnosis confirmed by at least two different serological tests for anti-Trypanosoma cruzi based on different principles or with different antigenic preparations, such as: enzyme-linked immunosorbent assay [ELISA], indirect immunofluorescence [IFI], indirect hemagglutination [IHA], western blot (WB), chemiluminescent immunoassay (CLIA). If documented history is not available, the tests may be performed during the screening

Key Exclusion Criteria:

* Patients with history of suspected or proven angioedema or unable to tolerate ACEIs, ARBs or ARNI (e.g., due to cough, hypotension, renal dysfunction, hyperkalemia)
* Use of sacubitril/valsartan in the past 3 months
* Patients requiring continuous intravenous inotropic therapy or with indication of advanced support intervention for HF:

  1. already on list for a heart transplantation
  2. with current indication of left ventricular assist device, or cardiac resynchronization therapy (CRT)
* Systemic systolic blood pressure lower than 95 mmHg or symptomatic hypotension
* Serum potassium > 5.2 mmol/L
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 of body surface area
* Severe gastrointestinal form of chronic Chagas' disease (demonstrated megaesophagus and/or important megacolon, e.g.: with compromised oral intake or surgical indication).
* Clinical conditions or systemic diseases limiting proper patient participation
* Pregnant or nursing women or women of child-bearing potential unless they are using highly effective methods of contraception
* Presence of other cardiac conditions:

  1. Previous cardiac surgery
  2. Heart failure where, in the Investigator's judgement, there is a possible alternative primary etiology e.g., due to coronary artery disease, valve disease, congenital heart disease or other causes.
  3. Untreated arrhythmia or serious conduction disease e.g., bradyarrhythmias, atrial fibrillation with rapid ventricular response, second or third degree atrioventricular block, etc.
  4. Primary uncorrected valvar pathology like moderate to severe aortic stenosis, mitral stenosis and primary mitral regurgitation
  5. Planned organ transplantation (or in listing for transplantation), planned cardiac or other major surgery (including ventricular assist device implantation)
* History of malignancy of any organ system within the past 5 years.
* Current confirmed COVID19 infection
* Past COVID19 infection with persistent symptom burden suspected due to COVID19 (persistent symptoms may include, but are not limited to, continued cough, breathing difficulty, muscle/joint aches, and gastrointestinal symptoms from the time of COVID19 infection onward)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 918 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Hierarchical composite endpoint composed of time to CV death, time to first HF hospitalization, relative change in NT-proBNP from baseline to Week 12 | Total follow up time up to approximately 36 months
  The primary efficacy endpoint will be analyzed using the win ratio approach comparing every participant in the sacubitril/valsartan arm to every participant in the enalapril arm to determine a winner. The estimated win ratio (the total number of winners in the sacubitril/valsartan arm divided by the total number of winners in the enalapril arm) will be provided. A winner in the pair-wise comparison has a delayed time to the occurrence of CV death; if time to the occurrence of CV death is censored, a winner has a delayed time to the occurrence of first HF hospitalization event; if the times to both CV events are censored, a winner has a more favorable (less increase or more decrease) change in NT-proBNP between Baseline and Week 12.

SECONDARY OUTCOMES:
Time to the first occurrence of a composite of CV events | From the date of randomization to the first occurrence (total follow up time up to approximately 36 months)
  Time from randomization to the first occurrence of HF hospitalization or CV death
Time to all-cause mortality | From date of randomization until the date of death from any cause assessed up to the end of the study, which is estimated to be up to approximately 36 months
  The time to all-cause mortality will be determined.
Time to sudden death or resuscitated sudden cardiac arrest | From date of randomization until the date of the sudden death or resuscitated sudden cardiac arrest assessed up to the end of the study, which is estimated to be up to approximately 36 months
  The time to sudden death or resuscitated sudden cardiac arrest will be determined.
Number of visits to an ER due to HF (where intravenous therapy is required) | From the date of randomization up to End of Study (EOS) assessment. Total follow up time up to approximately 36 months.
  The rate of visits to an emergency room (ER) due to HF (where intravenous therapy is required) will be determined.
Number of days alive out of the hospital | From the date of randomization up to End of Study (EOS) assessment. Total follow up time up to approximately 36 months.
  The number of days alive out of the hospital will be determined.
Number of ventricular fibrillation or sustained ventricular tachycardia | From the date of randomization up to End of Study (EOS) assessment. Total follow up time up to approximately 36 months.
  The number of ventricular fibrillation or sustained ventricular tachycardia needing specific pharmacological, electrical or other treatment will be determined.
Number of anti-tachycardia pacing or shock therapies | From the date of randomization up to End of Study (EOS) assessment. Total follow up time up to approximately 36 months.
  This will be determined in a subset on a subset of participants who have an ICD or CRT-D at Randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (56):
- Argentina (16):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, San Martín, Buenos Aires
  - Novartis Investigative Site, Temperley, Buenos Aires
  - Novartis Investigative Site, Villa María, Córdoba Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, San Miguel de Tucumán, San Miguel de Tucuman
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel Tucuman, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Formosa
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Santa Fe
  - Novartis Investigative Site, Santiago del Estero
- Brazil (30):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Brasila, Federal District
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, São Luís, Maranhão
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Montes Claros, Minas Gerais
  - Novartis Investigative Site, Passos, Minas Gerais
  - Novartis Investigative Site, Uberaba, Minas Gerais
  - Novartis Investigative Site, Uberlândia, Minas Gerais
  - Novartis Investigative Site, Londrina, Paraná
  - Novartis Investigative Site, Belém, Pará
  - Novartis Investigative Site, Recife, Pernambuco
  - Novartis Investigative Site, Teresina, Piauí
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Ijuí, Rio Grande do Sul
  - Novartis Investigative Site, Botucatu, São Paulo
  - Novartis Investigative Site, Bragança Paulista, São Paulo
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Indaiatuba, São Paulo
  - Novartis Investigative Site, Marília, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, Sao Jose Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Tatuí, São Paulo
  - Novartis Investigative Site, Votuporanga, São Paulo
  - Novartis Investigative Site, São Paulo
- Colombia (6):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Santa Marta, Magdalena Department
  - Novartis Investigative Site, San Gil, Santander Department
  - Novartis Investigative Site, Bogota DC
  - Novartis Investigative Site, Florida Blanca
  - Novartis Investigative Site, Floridablanca
- Mexico (4):
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, Ciudad de
  - Novartis Investigative Site, Oaxaca City
  - Novartis Investigative Site, Xalapa

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Lopes RD, Bocchi EA, Echeverria LE, Demacq C, de Barros E Silva PGM, Barbosa LM, Damiani L, Sayyed S, Yoshida LAF, Furtado RHM, Morillo CA, Kevorkian R, Ramires F, Bahit MC, Magana A, Chavez-Mendoza A, Miguel da Silva AH, Coelho da Silva A, Freitas AF Jr, Romano AA, Parneix A, Segura A, Franca CCB, Botta CE, de Barros E, Perna ER, Montenegro E, Quiroz Diaz FR, Feitosa-Filho GS, Severini GV, Molina I, Miranda JDSS, Sala J, Kerr Saraiva JF, Carbajales J, Maia LN, Santana Passos LC, Simoes MV, Moreira MDCV, Nunes MCP, Hernandes ME, Hominal M, Zarandon RS, Leon de la Fuente R, Aras R, Bazan SGZ, Luiz da Silva T Jr, Madrini V, de Oliveira WA Jr, Saporito WF, Gimpelewicz C, McMurray JJV; Prevention and Reduction of Adverse Outcomes in Chagasic Heart Failure Trial Evaluation (PARACHUTE-HF) Investigators. Sacubitril/Valsartan vs Enalapril in Heart Failure Due to Chagas Disease: An Open-Label, Multicenter Randomized Clinical Trial. JAMA. 2026 Jan 6;335(1):49-59. doi: 10.1001/jama.2025.19808. PMID 41335448
- [Derived] Bocchi EA, Echeverria LE, Demacq C, de Barros E Silva PGM, Mazza Barbosa L, Chiang LM, Damiani L, Morillo CA, Kevorkian R, Ramires F, Bahit MC, Ferrari A, Chavez-Mendoza A, Magana-Serrano JA, McMurray JJV, Gimpelewicz C, Lopes RD; PARACHUTE-HF Investigators. Sacubitril/Valsartan Versus Enalapril in Chronic Chagas Cardiomyopathy: Rationale and Design of the PARACHUTE-HF Trial. JACC Heart Fail. 2024 Aug;12(8):1473-1486. doi: 10.1016/j.jchf.2024.05.021. PMID 39111953